Date: 2025-08-31

**Unique Protocol ID: 2024-07566-01** 

Title: The Time Before the Crime - Risk Patterns in Offenders Undergoing a Forensic Psychiatric

**Evaluation (Tibec)** 

Principal Investigator: Katarina Howner, Associate professor, Karolinska Institutet

# **Review Template for Medical Record Review**

| Case Number (anonymize | d): | | |
|---|---|---|---|
| Gender: ☐ Male ☐ Fema | ale | | |
| Age at Index Offense: | | | |
| Age group: ☐ 18-24 years ☐ 25-39 years ☐ ≥ 40 years | | | |
| Unit(s) Reviewed: | | | |
| ☐ Outpatient only ☐ Inp | patient only Eme | rgency department only | ☐ Multiple units |
| Review Period: | | | |
| Review Performed By: | | | |
| Markers | | | |
| | 1 (15) | 0 1 11 1 (00) | - () |

| Marker | Inpatient (IP) | Outpatient (OP) | Emergency (ED) |
|---|---|---|---|
| Benzodiazepines or benzodiazepine-like medications | | | |
| Central stimulant medications | | | |
| Lack of treatment/intervention | | | |
| Non-adherence to treatment/intervention | | | |
| Compulsory psychiatric care | | | |
| Coercive measures | | | |
| Absence of violence risk assessment | | | |
| Increased psychiatric care needs | | | |
| Parallel psychiatric care contacts | | | |
| Polypharmacy (≥ 5 psychiatric meds) | | | |
| Weapon possession or interest | | | |

| Firearm unsuitability report |
|--------------------------------------|
| Suicide attempt |
| Historical suicide attempt |
| Aggression or violence |
| History of aggression or violence |
| Missed healthcare appointment |
| Missed appointment without follow-up |
| Multiple psychiatric diagnoses |
| Safeguarding concern report |
| Police transport to care |
| Substance use (excluding alcohol) |
| Alcohol use |
| Negative life event |
| Social vulnerability |
| Absence of crisis plan |

IP = Inpatient care, OP = Outpatient care, ED = Emergency department

#### **List of Markers with Definitions**

## Benzodiazepines or benzodiazepine-like medications

**Definition**: The marker is considered positive if the patient was prescribed or administered a benzodiazepine or a benzodiazepine-like medication during the review period.

Note: Benzodiazepine-like medications refer to the substances Zopiclone and Zolpidem

#### **Central stimulant medications**

**Definition**: The marker is considered positive if the patient was prescribed or administered central stimulant medications during the review period.

## Lack of treatment/intervention

**Definition**: The marker is considered positive if the patient had no treatment or intervention prescribed for their (main) diagnosis during the review period.

**Note**: Treatment refers to psychological or pharmacological treatment. Intervention refers to actions addressing issues resulting from diagnoses that do not primarily require pharmacological or psychological treatment (such as autism or intellectual disability), e.g., municipal housing, services under the LSS Act, or legal guardian.

If the patient lacks a main diagnosis, the diagnosis made at, e.g., an emergency visit is considered.

#### Non-adherence to treatment/intervention

**Definition**: The marker is considered positive if the patient was prescribed treatment or intervention but showed non-adherence during the review period.

**Note**: Non-adherence includes missed injections, low drug levels, failure to take medication, missed therapy appointments, not collecting medication from the pharmacy, or not residing in designated housing.

## Compulsory psychiatric care

**Definition**: The marker is considered positive if the patient was treated under the Compulsory Psychiatric Care Act or the Forensic Psychiatric Care Act at least once during the review period.

**Note**: It is also positive if a medical certificate about compulsory care was issued and a detention decision was made, even if no final commitment decision followed.

#### **Coercive measures**

**Definition**: The marker is considered positive if the patient was subject to coercive measures decided by the chief physician under the Compulsory Psychiatric Care Act or the Forensic Psychiatric Care Act during the review period.

#### Absence of violence risk assessment

**Definition**: The marker is considered positive if no documented violence risk assessment was made during psychiatric care visits within the review period.

Note: If an assessment exists, the marker is negative regardless of quality or risk rating.

#### Increased psychiatric care needs

**Definition**: The marker is positive if the patient had any of the following during the review period:

- a) ≥2 inpatient admissions,
- b) ≥1 readmission within one week after discharge,
- c) ≥2 emergency visits,
- d) ≥1 inpatient stay lasting over two months.

#### Parallel psychiatric care contacts

**Definition**: The marker is considered positive if the patient had parallel psychiatric care contacts with both general psychiatry and specialized addiction services.

**Note**: Includes outpatient visits, inpatient admissions, or emergency visits. Excludes municipal addiction care.

## Polypharmacy (≥ 5 psychiatric medications)

**Definition**: The marker is positive if the patient was prescribed ≥5 psychiatric medications at any point during the review period.

**Note**: Includes medications for psychiatric symptoms and narcotic substances like opioids and Pregabalin, both regular and PRN (when required).

## Weapon possession or interest

**Definition**: The marker is considered positive if the patient had access to weapons, carried a weapon during a search, or expressed current or historical interest in weapons during the review period.

**Note**: Weapons refer to firearms or knives.

## Firearm unsuitability report

**Definition**: The marker is considered positive if a report was filed with the police during the review period regarding the patient's unsuitability to possess firearms, in accordance with Chapter 6, Section 6 of the Swedish Firearms Act (1996:67).

## Suicide attempt

**Definition**: The marker is considered positive if the patient attempted suicide at least once during the review period.

**Note**: Includes all acts intended to end life. If intent is denied or unclear, it is still considered positive if the event required medical care.

#### Historical suicide attempt

**Definition**: The marker is considered positive if there is information indicating the patient attempted suicide at least once before the review period.

**Note**: Includes all acts intended to end life. If intent is denied or unclear, it is still considered positive if the event required medical care.

#### **Aggression or violence**

**Definition**: The marker is considered positive if the patient displayed aggressive or violent behavior toward objects, others, or self during the review period.

**Note**: Behavior must be documented as a clinical observation or from history. Includes all types of self-harm, e.g., cutting.

## History of aggression or violence

**Definition**: The marker is considered positive if there is information indicating the patient had shown aggressive or violent behavior before the review period.

**Note**: Behavior must be documented as a clinical observation or from history. Includes all types of self-harm, e.g., cutting.

## Missed healthcare appointment

**Definition**: The marker is considered positive if the patient missed or canceled at least one scheduled healthcare appointment during the review period.

#### Missed appointment without follow-up

**Definition**: The marker is considered positive if the patient missed or canceled at least one appointment during the review period without adequate follow-up by the healthcare provider.

**Note**: Adequate follow-up includes phone contact, home visits, or rescheduling.

#### Multiple psychiatric diagnoses

**Definition**: The marker is considered positive if the patient had psychiatric diagnoses from three or more different diagnostic clusters during the review period. Diagnoses must be recorded using ICD codes.

**Note**: Clusters are based on the first number following the F in ICD codes. For example, F20.3 and F29.9 are in the same cluster. An example of three different clusters: F20.0 (schizophrenia), F10.0 (alcohol intoxication), F84.1 (autism).

## Safeguarding concern report

**Definition**: The marker is considered positive if a family member or other person reported a concern about the patient's mental state to psychiatry, or if a report was made to social services in accordance with Chapter 14, Section 1 of the Social Services Act (2001:453).

## Police transport to care

**Definition**: The marker is considered positive if the patient arrived at psychiatric care with police assistance during the review period, either:

- a) voluntarily,
- b) under Section 11 of the Police Act (1984:387),
- c) under the Care of Intoxicated Persons Act (1976:511), or
- d) under Section 47 of the Compulsory Psychiatric Care Act (1991:1128).

## **Substance use (excluding alcohol)**

**Definition**: The marker is positive if the patient during the review period:

- a) had ≥1 substance use diagnosis,
- b) self-reported use,
- c) tested positive for non-prescribed narcotics,
- d) was reported to social services under the Care of Substance Abusers Act (1988:870), or
- e) was assessed by a physician according, Section 9 of the Care of Substance Abusers Act (1988:870).

Note: Alcohol use is excluded from this marker.

#### Alcohol use

**Definition**: The marker is positive if the patient during the review period:

- a) had ≥1 alcohol-related diagnosis,
- b) self-reported overuse,
- c) had >0.30 µmol/L phosphatidylethanol,
- d) was reported to social services under the Care of Substance Abusers Act (1988:870), or
- e) was assessed by a physician according, Section 9 of the Care of Substance Abusers Act (1988:870).

**Note**: This marker refers solely to alcohol use or dependence.

# **Negative life event**

**Definition**: The marker is considered positive if the patient experienced a negative life event (e.g., separation, bereavement, unemployment, or housing loss) during the review period and psychiatry was informed.

## **Social vulnerability**

**Definition**: The marker is considered positive if the patient was in a socially vulnerable situation that significantly affected functioning during the review period.

**Examples**: lack of social network, homelessness, or no source of income.

# Absence of crisis plan

**Definition**: The marker is considered positive if there was no crisis plan in the patient's record during the 12 months preceding the index offense date.

**Note**: This refers to the full year before the offense, not just the 3-month review period. The marker is positive only if the plan is entirely missing or older than 12 months.